CLINICAL TRIAL: NCT05400720
Title: Peer Support In Dialysis: A Feasibility Study
Brief Title: Peer Support In Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SIH131_Peer Mentoring
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-07

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: We aim to conduct the study over 6 to 12 months to obtain enough experience to enable feasibility evaluation.
  Mentor pool sample size: We anticipate having about 10 patients in the mentors' pool during the study period.
  Mentee sample size: We anticipate approaching between 20 to 30 dialysis patients over the study period.
  Supporting team: All members of the supporting staff will be invited to participate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mentee (Experimental): Participants will be approached by a mentor, exchange experiences and invite the prospective mentee to the program. Those interested to continue will undergo matching based on their desired criteria.
  Interventions: Behavioral: Mentoring

INTERVENTIONS:
Behavioral: Mentoring — At least one meeting between the mentor and mentee will occur to share experiences and see if the mentee would like to continue meeting with a mentor

SUMMARY:
Peer mentoring is an approach used to support patients through their experience. In the End Stage Kidney Disease community many patients find out about their kidney failure without warning. This study is designed to test the feasibility of a structured peer support program, specifically, patient uptake, engagement and patient and staff perspectives.

ELIGIBILITY:
Mentor Patient Participants Inclusion criteria:

* Patients living with dialysis or kidney transplant, who volunteer to support other patients.
* Mentor participants agree to complete the CMS End Stage Renal Disease Network Peer Mentoring training program (https://www.kidneylearninghub.com/patients-peer-mentoring-program/ ) and follow the guidelines for participation in the program.

Mentor Patient Participants Exclusion criteria:

* Age <18 years.
* Patient cannot communicate in English.
* Concerns raised by the clinical team that may expose the mentor, mentee, staff, or the program to risks, as identified by the clinical team and discussed with the principal investigator.

Mentee Patient Participants Inclusion criteria:

* All incident (new) dialysis patients or their care partners, within the first three months of dialysis.

OR

* Prevalent dialysis patients or their care partners identified by the clinical team to need peer support.

Mentee Patient Participants Exclusion criteria:

* Age < 18 years.
* Significant physical or psychological health conditions (including cognitive impairment) that would limit the patient's ability to interact with the mentor, AND care partner not available or reachable to join the program.
* This criteria will be subjectively evaluated by the clinical team.

Clinical and administrative staff supporting the program inclusion criteria

* referring physicians, the medical director of the center, social workers, nurses, patient care technicians (PCT), certified clinical hemodialysis technicians (CCHT), and administrative staff.
* Support staff are those who interact with mentors or mentees as part of their routine work.
* Formally participate in supporting the program by identifying candidates, introducing them to the program, or providing them with support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Mentor | 6 - 12 months
  Number of patients registering to become mentors, percent of those registered completing mentor training and percent of trained mentors who meet at least one mentee.
Mentee | 1 month
  Number and proportion of patients starting dialysis, or prevalent dialysis patients identified by the clinical team to need peer support, who receive an introductory peer mentor visit. Number and % of mentees who indicate interest to continue with more peer mentoring visits.

SECONDARY OUTCOMES:
Mentor Perspectives | 6-12month
  Evaluation of recruitment, training and program. Data collection will be through the Mentor Recruitment and Training Evaluation form and through focus group discussions
Mentee Perspectives | 1-4 weeks
  Peer Mentorship Program Evaluation - Mentee form to be completed by the mentee to collect data on the mentees perspective of the program
Support Staff Perspectives | 3,6,9 and 12 months
  Peer Mentorship Program Evaluation - Staff to be completed by the center staff to collect data on their perspective of the program
Mentor - Mentee Matching | 1 month
  Preferences about matching (n and % for age range, gender, race, language, social conditions, specific dialysis experiences [e.g. Peritoneal Dialysis / Home HemoDialysis / transplant], and others).

CONTACTS AND LOCATIONS:
Overall Officials: Wael Hussein, MD, Principal Investigator — Satellite Healthcare
Locations (2):
- United States (2):
  - Satellite Healthcare Mountain View, Mountain View, California
  - WellBound Mountain View, Mountain View, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett PN, St Clair Russell J, Atwal J, Brown L, Schiller B. Patient-to-patient peer mentor support in dialysis: Improving the patient experience. Semin Dial. 2018 Sep;31(5):455-461. doi: 10.1111/sdi.12703. Epub 2018 May 2. PMID 29722062
- [Background] Collins, K. (2016). NKF Peers Mentoring Program. National Kidney Foundation Journal of Nephrology Social Work, 40(2), 25-33.
- [Background] Fida'Husain, H. K., & Johan, A. (2020). Effects of Peer Support Program on Self-Management in Patients with End-Stage Renal Disease Undergoing Hemodialysis.
- [Background] Flythe JE, Narendra JH, Yule C, Manivannan S, Murphy S, Lee SD, Strigo TS, Peskoe S, Pendergast JF, Boulware LE, Green JA. Targeting Patient and Health System Barriers To Improve Rates of Hemodialysis Initiation with an Arteriovenous Access. Kidney360. 2021 Feb 26;2(4):708-720. doi: 10.34067/KID.0007812020. eCollection 2021 Apr 29. PMID 35373037
- [Background] Hussein WF, Bennett PN, Schiller B. Innovations to Increase Home Hemodialysis Utilization: The Transitional Care Unit. Adv Chronic Kidney Dis. 2021 Mar;28(2):178-183. doi: 10.1053/j.ackd.2021.02.009. PMID 34717865
- [Background] Orsmond GI, Cohn ES. The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions. OTJR (Thorofare N J). 2015 Jul;35(3):169-77. doi: 10.1177/1539449215578649. PMID 26594739
- [Background] St Clair Russell J, Southerland S, Huff ED, Thomson M, Meyer KB, Lynch JR. A Peer-to-Peer Mentoring Program for In-Center Hemodialysis: A Patient-Centered Quality Improvement Program. Nephrol Nurs J. 2017 Nov-Dec;44(6):481-496. PMID 29281772
- See also: Centers for Medicare and Medicaid Services (CMS). (2021). Partnership for patients. — https://partnershipforpatients.cms.gov/about-the-partnership/patient-and-family-engagement/the-patient-and-family-engagement.html
- See also: ESRD National Coordinating Center. (2021). ESRD Networks Peer Mentor Program. — https://esrdncc.org/en/patients/peer-mentoring-resources/
- See also: Lessons Learned: Implementation of a Peer-to-Peer Mentor Program in Individuals Requiring Hemodialysis. — http://dx.doi.org/10.37526/1526-744X.2021.48.4.399